# MC1841 / 18-003525

# Phase II Study of Niraparib and TSR-042 in Patients with Germline or Somatic BRCA1/2 and PALB2-related Pancreatic Cancer

NCT04493060

Document Date: 10/19/2023



Name and Clinic Number

Protocol #: MC1841 Version Date: 07Oct2023

# RESEARCH PARTICIPANT CONSENT AND PRIVACY AUTHORIZATION FORM

Study Title: MC1841: Phase II Study of Niraparib and TSR-042 in Patients with Germline or

Somatic BRCA1/2 and PALB2-related Pancreatic Cancer

**IRB#:** 18-003525

Principal Investigator: Dr. Robert McWilliams and Colleagues

# **Key Study Information**

This section provides a brief summary of the study. It is important for you to understand why

| the research is being done and what it will involve before you decide. Please take the time read the entire consent form carefully and talk to a member of the research team before making your decision. You should not sign this form if you have any questions that have not provided the research team before making your decision. |
|---|
| · · |
| · · |
| making your decision. Tou should not sign this form if you have any questions that have in |
| been answered. |
| This is a research study. Being in this research study is your choice; |
| you do not have to participate. If you decide to join, you can still sto |
| It's Your Choice at any time. You should only participate if you want to do so. You want to do so. |
| not lose any services, benefits or rights you would normally have if |
| you choose not to take part. |
| The purpose of this research is to further define genetic identification |
| of patients with your condition and to evaluate the treatment |
| combination of niraparib and dostarlimab (TSR-042) in patients wit |
| 1 , 1 |
| <b>Research Purpose</b> germline or somatic mutations in BRCA1/2 or PALB2. |
| You have been asked to take part in this research because you have |
| germline or somatic BRCA1/2 or PALB2-related pancreatic cancer. |

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



# Name and Clinic Number


| What's Involved | Study participation involves a combination treatment of two investigational drugs, niraparib and dostarlimab. Niraparib is an oral drug (pill form) that will be self-administered daily while on study. Dostarlimab is a drug that will be administered intravenously once at the beginning of each treatment cycle. Cycles are 21 days long and subjects will visit the clinic on Day 1 of each cycle (plus Day 15 of the first cycle). Subjects enrolled in this study will be asked to provide both blood samples (up to 6) and tissue samples (up to 2 biopsies with an optional |
|---|---|
| | 3 <sup>rd</sup> ) for research purposes at time points specified later in this form. The most common and expected risks of treatment with niraparib include low blood cell counts, high blood pressure, heart palpitations, urinary tract infection, shortness of breath, runny or stuffy nose, cough, headache, dizziness, feeling weak, lack of energy, difficulty sleeping, joint pain, back pain, stomach pain, indigestion, feeling sick, vomiting, watery stools (diarrhea), difficulty passing stool (constipation), and decreased appetite. |
| | The most common and expected risks of treatment with dostarlimab include anemia, nausea vomiting, diarrhea, itchy skin, rash, and increased levels in liver function tests. |
| Key Information | The risks of the tumor biopsy procedure are mainly pain, bleeding, and infection. Depending on the location of the tumor, there is a small risk of injury or damage to the nearby organs or tissues. Your doctor may use a local anesthetic and/or a medicine to calm your nerves before or during the biopsy procedure; there is a possibility that an allergic reaction to the anesthetic may occur. There is also a risk of scarring at the biopsy site, and there is a possibility of tumor cells spreading from the tumor into the nearby area. Your doctor will explain the procedure to you and discuss these risks with you. |
| | A complete, detailed list of any/all risks related to study participation is located later in this form in section "What are the possible risks or discomforts from being in this research study?" |

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


| | If you are interested in learning more about this study, read the rest of |
|---|---|
| | this form carefully. The information in this form will help you decide |
| Learn More | if you want to participate in this research or not. A member of our |
| | research team will talk with you about taking part in this study before |
| | you sign this form. If you have questions at any time, please ask us. |

# **Making Your Decision**

Taking part in research is your decision. Take your time to decide. Feel free to discuss the study with your family, friends, and healthcare provider before you make your decision. Taking part in this study is completely voluntary and you do not have to participate.

If you decide to take part in this research study, you will sign this consent form to show that you want to take part. We will give you either a printed or electronic copy of this form to keep. A copy of this form will be put in your medical record.

For purposes of this form, Mayo Clinic refers to Mayo Clinic in Arizona, Florida and Rochester, Minnesota; Mayo Clinic Health System; and all owned and affiliated clinics, hospitals, and entities.

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


# **Contact Information**

| If you have questions about | You can contact |
|---|---|
| <ul> <li>Study tests and procedures</li> </ul> | Principal Investigators: |
| <ul> <li>Materials you receive</li> </ul> | Robert McWilliams, MD (MN) |
| <ul> <li>Research-related appointments</li> <li>Research-related concern or complaint</li> </ul> | <b>Phone:</b> (507) 284-2511 |
| Research-related injuries or emergencies | Daniel Ahn, DO (AZ) |
| <ul> <li>Withdrawing from the research study</li> </ul> | <b>Phone:</b> (480) 301-8000 |
| | Hani Babiker, MD (FL) |
| | <b>Phone:</b> (904) 953-2000 |
| | Institution Name and Address: |
| | Mayo Clinic |
| | 200 1st Street SW |
| | Rochester, MN 55905 |
| | Mayo Clinic Hospital |
| | 5777 E. Mayo Boulevard |
| | Phoenix, AZ 85054 |
| | Mayo Clinic Florida |
| | 4500 San Pablo Road |
| | Jacksonville, FL 32224 |
| <ul><li>Rights of a research participant</li></ul> | Mayo Clinic Institutional Review Board (IRB) |
| | <b>Phone:</b> (507) 266-4000 |
| | <b>Toll-Free:</b> (866) 273-4681 |
| <ul> <li>Rights of a research participant</li> </ul> | Research Participant Advocate (RPA) |
| <ul> <li>Any research-related concern or complaint</li> </ul> | (The RPA is independent of the Study Team) |
| <ul> <li>Use of your Protected Health Information</li> </ul> | <b>Phone:</b> (507) 266-9372 |
| <ul> <li>Stopping your authorization to use your<br/>Protected Health Information</li> </ul> | <b>Toll-Free:</b> (866) 273-4681 |
| <ul> <li>Withdrawing from the research study</li> </ul> | E-mail: researchparticipantadvocate@mayo.edu |
| Billing or insurance related to this research | Patient Account Services |
| study | Toll-Free: (844) 217-9591 |

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



#### Name and Clinic Number


#### Other Information:

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# Why are you being asked to take part in this research study?

You are being asked to take part in this research study because you have germline or somatic BRCA1/2 and PALB2-related pancreatic cancer.

The plan is to have about 23 people take part in this study at Mayo Clinic.

# Why is this research study being done?

The purpose of this study is to further identify trends in the genetic information of patients with your condition and to evaluate the treatment combination of niraparib and dostarlimab (TSR-042) in patients with germline or somatic mutations in BRCA1/2 or PALB2.

# Information you should know

# Who is Funding the Study?

GlaxoSmithKline (GSK) is funding this study. GSK will pay Mayo Clinic to cover costs related to running the study.

#### **Information Regarding Conflict of Interest:**

Your healthcare provider may be referring you to this research study. If your healthcare provider is also an investigator on this study, there is the chance that his or her responsibilities for the study could influence his or her recommendation for your participation. If you prefer, your healthcare provider will be happy to refer you to another investigator on the research study team for you to decide if you want to participate in the study and to see you for the research study activities while you are in the study.

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


# How long will you be in this research study?

It will take you about 5-6 months to complete this research study. During this time, we will ask you to make 12-15 study visits to Mayo Clinic. However, if you are responding well to the study treatment, you may continue to remain on study until you decide to stop.

# What will happen to you while you are in this research study?

If you agree to be in the study, you will be asked to participate in the following:

# **Screening Visit**

During this visit, we will do some tests and procedures to see if you are eligible to take part in this research study. The Principal Investigator will review the results of these tests and procedures. If you aren't eligible, the Principal Investigator will tell you why. At this visit we will:

- Ask you about your medical history
- Give you a physical exam, including height, weight, and "vital signs" (blood pressure, temperature, heart and breathing rates)
- Draw a blood sample for clinical care testing
- Test your blood for pregnancy if you are able to become pregnant
- Ask you to provide a urine sample
- Conduct scan of your tumor (CT, MRI, or bone scan).

These exams, tests or procedures are part of regular clinical care and may be done even if you do not join the study. If you have had some of them recently, they may not need to be repeated. This will be up to the Principal Investigator.

<u>Study Treatment Visits</u> (every treatment cycle during this study is 21 days long)

# Cycle 1: Day 1

At this visit we will:

- Give you a physical exam, including measurements of your height, weight, and "vital signs" (blood pressure, temperature, heart and breathing rates)
- Ask you about any health problems since your last visit
- Provide you a medication diary for the oral study drug (niraparib)
- Provide a supply of the oral study drug and instructions for self-administration

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


Approval Date: October 19, 2023 Not to be used after: May 25, 2024

- Draw a blood sample for clinical care testing
- Test your blood for pregnancy if you are able to become pregnant
- Draw a blood sample for research
- Ask you to provide a urine sample
- Conduct a biopsy of your tumor
- Administer study drug (dostarlimab) intravenously

# Cycle 1: Day 8

- Ask you about any side effects or health problems since your last visit
- Draw a blood sample for clinical care testing

# Cycle 1: Day 15

At this visit we will:

- Ask you about any side effects or health problems since your last visit
- Draw a blood sample for research

# Cycle 2: Day 1 (and Day 1 of all remaining cycles)

At this visit we will:

- Give you a physical exam, including measurements of your weight and "vital signs" (blood pressure, temperature, heart and breathing rates)
- Ask you about any side effects or health problems since your last visit
- Review your medication diary
- Provide a supply of the oral study drug
- Draw a blood sample for clinical care testing
- Test your blood for pregnancy if you are able to become pregnant every third cycle after Cycle 1 (day 1 of Cycles 3, 6, 9, etc.)
- Draw a blood sample for research (Day 1 of Cycles 2, 3, 5 and last treatment visit only)
- Ask you to provide a urine sample
- Administer study drug (dostarlimab) intravenously
- Conduct scan of your tumor (CT, MRI, or bone scan). These scans will be done every 6 weeks starting with your screening visit (Day 1 of Cycles 2, 4, 6, etc.).
- Conduct a biopsy of your tumor (Day 1 of Cycle 5 and last treatment visit only; biopsy conducted during last treatment visit is optional)

#### Clinical Follow-up Visit (approximately 30 days after last treatment visit)

At this visit we will:

- Give you a physical exam, including measurements of your weight and "vital signs" (blood pressure, temperature, heart and breathing rates)
- Ask you about any side effects or health problems since your last visit

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


- Draw a blood sample for clinical care testing
- Test your blood for pregnancy if you are able to become pregnant
- Ask you to provide a urine sample

# **Event Monitoring Visits**

These visits will begin 3 months after the Clinical Follow-up Visit and will occur every three months after. During these visits, we will ask you about any health problems since your last visit.

# **Blood Pressure and Heart Rate Monitoring**

During the first 8 weeks of study treatment, you will be asked to monitor your blood pressure and heart rate at least once a week. You will be provided a diary for recording your blood pressure and heart and you will be asked to record those values at the beginning of each week (Days 1, 8, and 15 of Cycles 1, 2, and 3). If you are in the clinic for a study visit during any of those days, your blood pressure and heart rate will be recorded by the study staff and you will not have to record it in your diary.

#### **Collection of Blood and Tissue Samples for Research**

Tissue and blood specimens are mandatory for this study. You will be asked to have biopsies to collect tissue, and blood draws (taken at the same times as your clinical blood tests) for this study.

You will be informed of any clinically relevant research results. Any results reported to you individually, will also be placed in your medical record. Study results will be reported on ClinicalTrials.gov after the study is completed.

#### **Birth Control Requirements**

If you are sexually active and able to become pregnant, or able to cause pregnancy of someone able to become pregnant, you must agree to use one of the birth control methods listed below:

- Hormonal methods, such as birth control pills, patches, injections, vaginal ring, or implants
- Barrier methods (such as a condom or diaphragm) used with a spermicide (a foam, cream, or gel that kills sperm)
- Intrauterine device (IUD)
- Abstinence (no sex)

If you are of childbearing potential, you must use birth control for the entire study and for at least 180 days after your last dose of Niraparib and 180 days after your last dose of dostarlimab.

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


If you are a male subject and are sexually active with a person of childbearing potential, you must use birth control for the entire study and for at least 180 days after your last dose of Niraparib and 180 days after your last dose of dostarlimab.

If you are already using a method of birth control, your Study Doctor or the study staff will discuss with you whether your current method of birth control is acceptable for use during this study.

# What are the possible risks or discomforts from being in this research study?

#### Niraparib (Formerly MK-4827)

Niraparib has moderate influence on the ability to drive or use machines. Patients who take niraparib may experience weakness, fatigue, difficulty concentrating and dizziness. Patients who experience these symptoms should observe caution when driving or using machines.

Known side effects of niraparib are listed below:

#### Very Common occurrence (may affect more than 1 in 10 people)

- Decrease in a type of blood cell called platelets that help stop bleeding; this may increase your risk of bleeding (thrombocytopenia)
- Decrease in red blood cells that carry oxygen; this may make you feel tired or short of breath (anemia)
- Decrease in a type of white blood cell called a leukocyte that fight infection; this may decrease your ability to fight infections (leukopenia)
- Decrease in a type of white blood cell called neutrophils that fight infection; this may decrease your ability to fight infections and may be associated with fever, and may lead to a potentially life-threatening condition caused by the body's response to an infection, triggering changes that can damage multiple organ systems (neutropenia, febrile neutropenia)
- Increased blood pressure (hypertension)
- Noticeably rapid, strong, or irregular heartbeat (palpitations)
- Pain or burning when urinating which may indicate an infection (urinary tract infection)
- Breathlessness or difficulty breathing (dyspnea)
- Runny or stuffy nose (nasopharyngitis)
- Cough
- Headache
- Feeling lightheaded or like you are about to faint (dizziness)

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


- Feeling weak (asthenia)
- Feeling tired, lack of energy (fatigue)
- Sleeplessness, trouble sleeping (insomnia)
- Joint pain (arthralgia)
- Back pain
- Pain in your belly (abdominal pain)
- Indigestion (dyspepsia)
- Feeling sick to your stomach (nausea)
- Vomiting
- Frequent watery stools (diarrhea)
- Difficulty with emptying the bowels, often because of hard stools (constipation)
- Reduced desire to eat (decreased appetite)

# Common occurrence (may affect up to 1 in 10 people)

- Infection due to low white blood cell counts (neutropenic infection)
- Low blood cell counts due to a problem in the bone marrow or blood cancer starting from the bone marrow (Myelodysplastic Syndrome [MDS]/Acute Myeloid Leukemia [AML])
- An irritation or infection in the tubes that carry air in and out of the lungs, that causes a cough (bronchitis)
- An abnormally rapid heart rate (tachycardia)
- An accumulation of fluid that causes swelling in lower extremities such as lower legs, hands and feet (peripheral edema)
- Muscle pain (myalgia)
- Rash
- Decrease in weight
- Feelings of sadness, depressed (depression)
- Feelings of worry, nervousness, or unease (anxiety)
- Impaired concentration, understanding, memory, and thinking (cognitive impairment)
- Inflammation of the white area of the eye (conjunctivitis)
- Nosebleed (epistaxis)
- Sore, red mouth (stomatitis)
- Swelling or irritation of the lining of the mouth, throat, esophagus, stomach, or intestines (mucosal inflammation/mucositis)
- Abnormal taste in mouth (dysgeusia)
- Dry mouth
- Increased sensitivity of the skin to sunlight (photosensitivity)
- Decrease in levels of potassium in your blood (hypokalemia)
- Increased level of creatinine in your blood; this may be a sign of kidney damage (blood creatinine increase)

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


- Increased liver enzymes in the blood; aspartate transaminase ("AST"), alanine aminotransferase ("ALT"), gamma glutamyl transferase increased ("GGT"), or alkaline phosphatase (ALP); this may be a sign of damage to liver cells
- Allergic reaction (hypersensitivity, including anaphylaxis)

# **Uncommon Occurrence (may affect up to 1 in 100 people)**

- Fever with low white blood cell count (febrile neutropenia)
- Severe life-threatening infection due to low white cell counts [associated with low blood pressure and possible organ failure (for example, heart, kidney and/or liver)] (neutropenic sepsis)
- Decrease in number of all types of blood cells (pancytopenia)
- Confusion (confusional state/disorientation)
- Seeing or hearing things that are not really there (hallucination)
- Inflammation of the lungs which can cause shortness of breath and difficulty breathing (non-infectious pneumonitis)

# Rare Occurrence (may affect up to 1 in 1000 people)

- Severe increase in blood pressure (hypertensive crisis)
- A brain condition with symptoms including seizures, headache, confusion, and changes in vision (posterior reversible encephalopathy syndrome [PRES])

#### **Side Effects Requiring Immediate Medical Attention:**

The side effects listed below require IMMEDIATE MEDICAL ATTENTION OR ADVICE. Call the study staff right away if you have any of these side effects:

- Allergic reactions can be life-threatening. Symptoms may include difficulty breathing, shortness of breath, low blood pressure (feeling lightheaded, dizziness), tingling around the mouth, rash.
- Low platelet counts may increase your risk of bleeding and bruising. Bleeding may require urgent medical attention, including a transfusion (receiving blood or blood products by vein).
- Low red blood cell counts may make you feel tired or short of breath and symptoms may require a blood transfusion.
- Low neutrophil counts may be associated with infection, sometimes severe and life-threatening (neutropenic infection, neutropenic sepsis):
  - Symptoms of severe life-threatening infection may include fever, feeling of low blood pressure (lightheadedness, dizziness), decreased urination, rapid pulse, rapid breathing or shortness of breath
- Decrease in the number of all types of blood cells (pancytopenia)
- Low blood cell counts due to a problem in the bone marrow or blood cancer starting from the bone marrow (MDS or AML). MDS/AML, including fatal cases, have been reported

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


with use of niraparib. If you experience prolonged haematological toxicities, contact your study doctor for haematologist evaluation.

- High blood pressure (hypertension) including severe increase in blood pressure (hypertensive crisis) has been reported with the use of niraparib. If you have pre-existing hypertension, the physician will determine if your blood pressure is adequately controlled before starting niraparib treatment.
  - Symptoms of a severe increase in blood pressure may include blurry vision, headache, nausea, vomiting, confusion, passing out, seizures, weakness or numbness on one side of body or in one arm or leg and/or difficulty talking (symptoms of a stroke), trouble breathing, chest pain, pain in the upper or lower back, urine that is brown or bloody
- Posterior Reversible Encephalopathy Syndrome (PRES), a rare neurological side effect has been reported with niraparib treatment.
  - o If you have headache, vision changes, confusion or seizure with or without high blood pressure, please contact your doctor.

#### **Class Effects:**

Class effects are potential risks that are associated with a particular group of drugs. Niraparib belongs to the group known as poly (ADP-ribose) polymerase inhibitors (PARP) inhibitors. These class effects are potential risks for the group of drugs but have not yet been identified as side effects for niraparib.

#### Secondary Primary Malignancy:

PARP inhibitors may also cause a new primary cancer (that is, a cancer other than the one for which you have been treated). In 2 studies comparing niraparib to placebo (sugar pill), new primary cancers were observed in a small number of patients who took niraparib or placebo.

#### Safe Handling:

Niraparib may have adverse effects on an unborn baby. Wash your hands after handling the Study Drug. If a caregiver is giving the Study Drug to you, he or she should wear disposable gloves. Notify your Study Doctor if it appears that the Study Drug is damaged or defective in any way.

# **Dostarlimab (TSR-042)**

As of April 2023, dostarlimab has been studied in about 3000 patients with advanced or recurrent solid tumors in clinical trials, with about 2300 of these patients receiving dostarlimab in combination with other medicines Your study doctor will explain the risks, side effects, and discomforts that may be experienced related to non-study drugs which are part of usual care. Some of the side effects mentioned below can be life-threatening or fatal.

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


These side effects are considered <u>very common</u> in patients who took dostarlimab (may affect more than 1 in 10 people):

- Decrease in the number of red blood cells that carry oxygen. Low red blood cell count may make you feel tired or short of breath and symptoms may require a blood transfusion (anemia)
- Feeling sick to the stomach (nausea)
- Vomiting
- Frequent watery stools (diarrhea)
- Itchy skin (pruritus)
- Rash
- Fever (pyrexia)
- Increased levels of substances in the blood produced by the liver which may be a sign of liver injury (AST increased, ALT increased) (transaminases increased)
- Underactive thyroid gland (hypothyroidism)

These side effects are considered **common** in patients who took dostarlimab (may affect up to 1 in 10 people):

- Decreased production of adrenal hormones resulting in possible weakness and/or low blood pressure (adrenal insufficiency)
- Muscle pain (myalgia)
- Overactive thyroid gland (hyperthyroidism)
- Inflammation of the lungs which can cause shortness of breath and difficulty breathing (pneumonitis)
- Inflammation of the pancreas causing pain in the upper abdomen. This could become severe and cause nausea and vomiting, fever, and rapid heart rate (pancreatitis)
- Inflammation of the colon that can cause stomach pain or diarrhea (colitis)
- Chills
- Inflammation of the liver (hepatitis)

These side effects are considered <u>uncommon</u> in patients who took dostarlimab (may affect up to 1 in 100 people):

- Destruction of red blood cells which can cause tiredness, dizziness, yellow skin or fast heart rate (autoimmune hemolytic anemia)
- Inflammation of the thyroid gland (thyroiditis)
- Pituitary gland inflammation (hypophysitis)
- Severe high blood sugar due to uncontrolled diabetes (diabetic ketoacidosis)
- Diabetes requiring insulin (Type 1 diabetes mellitus)
- Inflammation of the eye which can cause redness, blurred vision or vision loss (uveitis)
- Muscle pain involving several muscles (polymyalgia rheumatica)

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


- Kidney inflammation (nephritis)
- Immune-mediated arthritis
- Myasthenia gravis
- Inflammation in the brain (encephalitis)
- Inflammation of the heart muscle (myocarditis)
- Inflammation of the lining of the stomach (gastritis)
- Inflammation of the food pipe (esophagitis)
- Inflammation of the small intestine (enteritis)
- Inflammation of blood vessels in the gastrointestinal tract (vasculitis gastrointestinal)
- Inflammation of the muscle which can cause weakness, swelling and pain (myositis)
- Inflammation throughout the whole body leading to high or low temperatures, low blood pressure, increased heart rate, increased rate of breathing and low or high white blood cell count (Systemic Inflammatory Response Syndrome)
- Infusion-related reactions which can occur within 24 hours after receiving an intravenous infusion, or which can be delayed for up to about 2 weeks. Infusion-related reactions may include dizziness or fainting, flushing, rash, fever, chills, shortness of breath, increased or decreased blood pressure, increased heart rate, swelling of the lips, tongue or face, feeling sick to your stomach, back pain or pain at the site of infusion. Although infusion-related reactions are usually reversible, they can be severe or life threatening. (Infusion related reactions)

There are rare but serious immune-related adverse events which have been seen when dostarlimab was used alone or in combination with other medicines:

- Overactive immune-system cells which damage body tissues and organs leading to signs of uncontrolled fever, enlarged spleen, low blood count and liver test abnormalities. This disease can be fatal. (Hemophagocytic Lymphohistiocytosis).
- A neurological disorder where the immune system attacks part of the peripheral nervous system that can cause tingling in the feet and hands, pain, muscle weakness, and problems with coordination (Guillain-Barre syndrome).
- Muscle weakness, twitching, cramping, or inability to move (peripheral motor neuropathy)
- Muscle pain and weakness; swollen, red, or thickened skin (eosinophilic fasciitis)

There may be other risks called "class effects" that have been seen in patients receiving other drugs that work like dostarlimab. These effects could also occur with dostarlimab. They are potential risks but not known as side effects for dostarlimab so far. The most significant class related side effects are "immune-related", meaning side effects caused by increased activity of the immune system, which can affect multiple organs of the body including bowels (gastrointestinal tract), hormone glands (endocrine system), heart (cardiovascular system), lungs,

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


liver, skin, muscles and joints (musculoskeletal system), and nerves (nervous system). These other immune-related side effects may be life-threatening or fatal.

The side effects listed below require <u>immediate medical attention or advice</u>. Call the study doctor right away if you have any of these side effects.

- Respiratory: shortness of breath, rapid breathing, new or worse cough
- Gastrointestinal: diarrhea, stools that are black or bloody, stomach area pain, nausea or vomiting
- Kidneys: dark or bloody urine, urinating more often than usual
- Musculoskeletal: chest pain, muscle pain or weakness
- Cardiac: fast or unusual heartbeat
- Skin: rash, itching, blisters, pale or yellow skin
- Eyes: yellowing of the whites of your eyes, blurry vision
- Brain: abnormal thinking, confusion, personality changes, headache and neck stiffness.
- General: bleeding or bruising more easily than normal, feeling cold, hair loss, dizziness or fainting, feeling tired or weak, fever or chills.

#### Risks related to pregnancy and breastfeeding

Dostarlimab may cause harm to the unborn baby when it is used by a pregnant person. You should not join this study if you are pregnant or planning to become pregnant. You should not join this study if you are breastfeeding.

If you are a woman able to have children, you will be given a pregnancy test at screening, and if the result is positive, you will not be able to participate in this study.

You will be required to use one highly effective form of contraception with your partner starting with the Screening Visit through 180 days after the last dose of study therapy. If you are already using a method of birth control, your Study Doctor or the study staff will discuss with you whether your current method of birth control is acceptable for use during this study.

The following are considered highly effective forms of contraception: hormonal contraceptives that include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents), intrauterine device (IUD), vasectomized partner, and abstinence, if this is the established and preferred contraception for the patient.

If, during this study, you or your partner become pregnant or think you may be pregnant, stop taking the Study Drug and let the Study Doctor know right away. You will be asked to withdraw from the study. Information about your pregnancy and its outcome will be collected and used to

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



#### Name and Clinic Number


learn more about the effects of the Study Drug on pregnancy. Payment for all aspects of obstetrical care, child, or related care will be your responsibility.

Female study participants who are pregnant or breast-feeding, or any study participant unable or unwilling to use effective contraception as required by study instructions should not use dostarlimab.

All drugs have a potential risk of an allergic reaction, which if not treated promptly, could become life-threatening.

Other less common side effects have been reported. The Study Doctor or staff can discuss these with you.

#### **Reproductive Risks**

The effect of the combination of niraparib and dostarlimab on a fetus (developing baby still in the womb), or on a breastfeeding infant, is unknown and may be harmful. Because of these risks, persons of childbearing potential cannot take part in this study if they are pregnant or breastfeeding.

Subjects of Childbearing Potential:

If you are able to become pregnant, you must have a negative pregnancy test in order to participate in this study unless you cannot become pregnant.

To participate in the study, patients who can become pregnant must adhere to the birth control requirements.

If you become pregnant or think you may be pregnant during the study, you must stop taking the study drugs and contact the Study Doctor's site **right away**. You will be asked to withdraw from the study. The Study Doctor is required to follow up and document the course and the outcome of all pregnancies, even if you withdraw from the study or if the study has finished.

You must not breast-feed an infant (or store breastmilk for use) during the study and for 90 days after receiving the final dose of Niraparib and for 180 days after receiving the final dose of dostarlimab.

Subjects Able to Father a Child:

To participate in the study, male study patients must adhere to contraception requirements.

You must not donate sperm for 180days after your last dose of Study Drug: If your partner thinks they might have become pregnant within one month of beginning the study, while you are in the study, or for 180 days after your last dose of dostarlimab or 180 days

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


after your last dose of niraparib, you must tell the Principal Investigator immediately. The Principal Investigator may ask for your partner's permission to collect information about the outcome of the pregnancy and the newborn. You won't have to stop taking the study drug or stop taking part in the study if your partner becomes pregnant.

#### **Other Risks**

#### **Blood Draw Risks**

The risks of drawing blood include pain, bruising, lightheadedness, and/or fainting, or rarely, infection at the site of the needle stick.

#### **MRI Risks**

There is no radiation associated with MRI, but people who have metal devices like pacemakers cannot have an MRI and will not be able to participate in the study. Some people with claustrophobia may feel too closed in and may not tolerate MRI scanning. If you feel too confined in the MRI scanner you can inform the technologist and the MRI scan will be stopped. The MRI machine makes loud knocking sounds when it is scanning. Because of this you will be asked to wear earplugs while getting your MRI scan. The earplugs minimize discomfort from noise and keep the MRI noise within the safety range.

The contrast agent you will receive is FDA-approved and used routinely for MRI exams. It contains a material called gadolinium, a rare metal. About 1 in 100 people may notice discomfort, tingling or warmth in the lips, metallic taste in the mouth, tingling in the arm, nausea, or headache. These side effects usually last only for a short time and go away as your body adjusts to the gadolinium. There is a small risk of an allergic reaction to gadolinium. However, a severe allergic reaction occurs in less than one in 300,000 people. The needle placed in your vein to give you the gadolinium may cause minor pain, bruising and/or infection at the injection site. Studies have shown that small amounts of gadolinium may remain in the body of patients who have received these injections. The effect of this, if anything, is unknown at this time.

#### **Radiation Risk**

You will be exposed to radiation from the CT scans of your tumor. The amount of radiation has a low risk of harmful effects.

#### **Biopsy Risks**

The risks of the tumor biopsy procedure are mainly pain, bleeding, and infection. Depending on the location of the tumor, there is a small risk of injury or damage to the nearby organs or tissues. Your doctor may use a local anesthetic and/or a medicine to calm your nerves before or during the biopsy procedure; there is a possibility that an allergic reaction to the anesthetic may occur.

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


There is also a risk of scarring at the biopsy site, and there is a possibility of tumor cells spreading from the tumor into the nearby area. Your doctor will explain the procedure to you and discuss these risks with you.

Complications from biopsies can be life threatening. As with any interventional procedure, other potentially serious complications from bleeding or organ damage may occur. These might require additional surgical intervention.

The risks described above may be different for you depending on your health and the location of the tumor. These risks should be discussed with your study doctor or person performing the biopsy.

You will be exposed to radiation during the CT-guided biopsies. The amount of radiation has a low risk of harmful effects.

#### **Bone and Bone Marrow Sample**

If your doctor wants you to be tested for Myelodysplastic Syndrome and Acute Myeloid Leukemia (MDS/AML), then you will have a bone/bone marrow biopsy collected for testing by a local haematologist. Your local haematologist may ask you to sign another consent form before the procedure. This procedure may take about 30 minutes, including the preparation of the biopsy site. Before the procedure, you will be given local anaesthesia or IV sedation (to numb the place where the biopsy will be taken). A needle will be placed either into your breastbone or a pelvic bone to obtain the liquid bone marrow sample. A second sample will be also collected by removing a small piece of the bone along with the marrow inside the bone. The doctor will be sure that you have recovered from the anaesthesia before you leave the doctor's office. Risks of the procedure may include a brief sharp pain during the procedure, bleeding (if you have low platelets (blood cells)), infection or discomfort at the site of biopsy.

#### **Genetic Testing Risks**

This study involves testing your DNA, which is the genetic information you inherited from your parents (also known as genetic testing). You will not be notified of the genetic test results and they will not be put into your medical record.

A Federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


• Employers with 15 or more employees may not use your genetic information when making a decision to hire, promote, or fire you or when setting the terms of your employment.

All health insurance companies and group health plans must follow this law.

Be aware that this new Federal law doesn't protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance.

#### **Standard of Care Risks**

Your doctor will discuss the risks of tests and procedures that are part of your standard clinical care.

# **Confidentiality Risk**

As with all research, there is a chance that confidentiality could be compromised; however, we take precautions to minimize this risk.

#### **Additional Costs**

Taking part in this research study may lead to added costs to you. In some cases, insurance will not pay for services ordinarily covered because these services were performed in a research study. You should check with your insurance company to see what services will be covered and what you will be responsible to pay.

#### **Unknown Risks**

There may be other side effects or risks that we cannot predict. Many side effects may go away shortly after the study medication or procedure is stopped. However, in some cases they can be serious, long-lasting, permanent, and/or fatal.

# Are there reasons you might leave this research study early?

If you decide to stop taking part in the study for any reason, we will ask you to make a final study visit. At this visit, we will:

- Ask you about side effects or health problems since your last visit
- Draw a blood sample for research
- Review your study drug diary
- Collect any unused study drug

You may decide to stop at any time. You should tell the Principal Investigator if you decide to stop and you will be advised whether any additional tests may need to be done for your safety.

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


In addition, the Principal Investigator or Mayo Clinic may stop you from taking part in this study at any time:

- if it is in your best interest,
- if you don't follow the study procedures,
- if the study is stopped.

If you leave this research study early, or are withdrawn from the study, no more information about you will be collected; however, information already collected about you in the study may continue to be used.

We will tell you about any new information that may affect your willingness to stay in the research study.

# What if you are injured from your participation in this research study?

#### Where to get help:

If you think you have suffered a research-related injury, you should promptly notify the Principal Investigator listed in the Contact Information at the beginning of this form. Mayo Clinic will offer care for research-related injuries, including first aid, emergency treatment and follow-up care as needed.

#### Who will pay for the treatment of research related injuries?

Care for such research-related injuries will be billed in the ordinary manner, to you or your insurance. Treatment costs for research-related injuries not covered by your insurance will be paid by Mayo Clinic.

# What are the possible benefits from being in this research study?

Others with pancreatic cancer may benefit in the future from what we learn in this research study.

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


# What alternative do you have if you choose not to participate in this research study?

You don't have to be in this study to receive treatment for your condition. For example:

- You may choose to try another treatment option determined by your doctor.
- You may choose to take part in a different study, if one is available.
- You choose not to receive treatment.

For patients who have only had one prior line of therapy for pancreatic cancer, there are other chemotherapy regimens with demonstrated benefit for second line treatment. You and your oncologist should discuss pros and cons to these alternatives.

Talk to the Principal Investigator or your doctor if you have any questions about any of these treatments or procedures.

# What tests or procedures will you need to pay for if you take part in this research study?

You won't need to pay for tests and procedures which are done just for this research study. These tests and procedures are:

- Supply and administration of the study drugs (niraparib and dostarlimab)
- Collection and testing of blood samples for research
- Collection and testing of tissue samples for research

However, you and/or your insurance will need to pay for all other tests and procedures that you would have as part of your clinical care. These tests and procedures are:

- Physical exams and health assessments (including blood tests conducted as part of your clinical care)
- Scans of your tumor (CT, MRI, or bone scans)
- Pregnancy testing

You will also be responsible for any co-payments and deductibles.

If you have billing or insurance questions call Patient Account Services at the telephone number provided in the Contact Information section of this form.

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



| Name and Clinic Number |
|------------------------|

# Will you be paid for taking part in this research study?

You won't be paid for taking part in this study.

There is a very small chance that some commercial value may result from the use of your sample. This could include new products like a drug or a test to diagnose a disease. If that happens, you will not be offered a share in any profits.

# Will your information or samples be used for future research?

Blood and tissue samples will be used for research related to the study and study drug. These samples may be analyzed at Mayo Clinic or sent externally to complete the testing. Research results will not be returned to you.

We would also like to keep your sample for future research. You can still take part in this current study even if you don't want your sample used for future research. If you agree to give your sample, it will be the property of Mayo Clinic.

Other researchers at Mayo Clinic who aren't involved with this study may ask to use your sample for future research. Researchers at other institutions may also ask for a part of your sample for future studies. If you approve release of your sample by checking 'yes' below, Mayo may send the sample(s) and some information about you to researchers who request them, but Mayo will <u>not</u> send your name, address, phone number, social security number, or any other identifying information with the sample. Your sample will be sent to researchers in a coded format, which protects your identity.

Some future studies may examine your DNA, which is the genetic information you inherited from your parents (genetic testing). The Principal Investigator may contact you if there are findings which may be useful for your health care. You would be given general information on the potential risks, benefits, and costs of choosing to learn about the findings.

# Please read the following statements and mark your choices:

| 1. I p | ermit my sample | to be stored and used in fut | cure research of pancreatic cancer at Mayo |
|---|---|---|---|
| Clinic | <b>:</b> | | |
| Yes | ☐ No | Please initial here: | Date: |

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number

Protocol #: MC1841
Version Date: 07Oct2023

Approval Date: October 19, 2023 Not to be used after: May 25, 2024

| | 2. I permit my sample to be stored and used in future research at Mayo Clinic to learn about, prevent, or treat any other health problems: | | | |
|---|---|---|---|---|
| | Yes | ☐ No | Please initial here: | |
| | 3. I permit Mayo Clinic to give my sample and related information to researchers at other institutions: | | | |
| | Yes | ☐ No | Please initial here: | |
| | 4. I permit Mayo Clinic to conduct an additional biopsy at the end of study treatment to collect tissue for research testing purposes: | | | |
| | Yes | ☐ No | Please initial here: | _Date: |
| Optional Research Biopsy If your cancer returns, we would like to obtain a portion of the biopsy tissue for research testing. These tests will be done in order to understand how your cancer responds to treatment. It is noted that this will help investigators better understand how to make this therapy more effective. The results of these tests will not be sent to you or your study doctor and will not be used in planning your care. These tests are for research purposes only, and you will not have to pay for them. | | | | |
| You can take part in the treatment portion of this study without taking part in these research aboratory tests. | | | | |
| 5. If my cancer comes back, I agree to an additional, optional biopsy to provide tissue sample(s) from my biopsy to Mayo Clinic for research testing planned as part of this study. | | | | |
| | Yes | ☐ No | Please initial here: | _Date: |
| There is a very small chance that some commercial value may result from the use of your donated sample. If that happens, you won't be offered a share in any profits. | | | | |
| You may request to have your sample destroyed by writing to the Principal Investigator. | | | | |

You may request to have your sample destroyed by writing to the Principal Investigator. The address is found in the "Contact Information" section of this consent form.

Your information and/or samples would be removed from any repository where they are stored, if possible. Information and/or samples already distributed for research use will not be retrieved. Because we cannot predict how your sample will be used in the future, we cannot promise that samples can be retrieved and destroyed.

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


# How will your privacy and the confidentiality of your records be protected?

Mayo Clinic is committed to protecting the confidentiality of information obtained about you in connection with this research study. All of your research samples will be labeled with a code number and kept in locked storage.

Only your study doctor will be able to link your samples with your identity. No one working with your samples will know your identity. If the results of the research are made public, information that identifies you will not be used.

During this research, information about your health will be collected. Under Federal law called the Privacy Rule, health information is private. However, there are exceptions to this rule, and you should know who may be able to see, use and share your health information for research and why they may need to do so. Information about you and your health cannot be used in this research study without your written permission. If you sign this form, it will provide that permission (or "authorization") to Mayo Clinic.

# Your health information may be collected from:

- Past, present and future medical records.
- Research procedures, including research office visits, tests, interviews and questionnaires.

# Your health information will be used and/or given to others to:

- Do the research.
- Report the results.
- See if the research was conducted following the approved study plan, and applicable rules and regulations.

# Your health information may be used and shared with:

- Mayo Clinic research staff involved in this study.
- Other Mayo Clinic staff involved in your clinical care.
- Researchers involved in this study at other institutions.
- The sponsor(s) of this study and the people or groups hired by the sponsor(s) to help perform this research.
- The Mayo Clinic Institutional Review Board that oversees the research.

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


- Federal and State agencies (such as the Food and Drug Administration, the Department of Health and Human Services, the National Institutes of Health and other United States agencies) or government agencies in other countries that oversee or review research.
- A group that oversees the data (study information) and safety of this research.

# How your information may be shared with others:

While taking part in this study, you will be assigned a code that is unique to you, but does not include information that directly identifies you. This code will be used if your study information is sent outside of Mayo Clinic. The groups or individuals who receive your coded information will use it only for the purposes described in this consent form.

If the results of this study are made public (for example, through scientific meetings, reports or media) information that identifies you will not be used.

In addition, individuals involved in study oversight and <u>not</u> employed by Mayo Clinic may be allowed to review your health information included in past, present, and future medical and/or research records. This review may be done on-site at Mayo Clinic or remotely (from an off-site location). These records contain information that directly identifies you. However, the individuals will not be allowed to record, print, copy (using paper, digital, photographic or other methods), or remove your identifying information from Mayo Clinic.

#### Is your health information protected after it has been shared with others?

Mayo Clinic asks anyone who receives your health information from us to protect your privacy; however, once your information is shared outside Mayo Clinic, we cannot promise that it will remain private and it may no longer be protected by the Privacy Rule.

# **Your Rights and Permissions**

Participation in this study is completely voluntary. You have the right not to participate at all. Even if you decide to be part of the study now, you may change your mind and stop at any time. You do not have to sign this form, but if you do not, you cannot take part in this research study.

Deciding not to participate or choosing to leave the study will not result in any penalty. Saying 'no' will not harm your relationship with your own doctors or with Mayo Clinic.

If you cancel your permission for Mayo Clinic to use or share your health information, your participation in this study will end and no more information about you will be collected; however, information already collected about you in the study may continue to be used.

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



Name and Clinic Number


You can cancel your permission for Mayo Clinic to use or share your health information at any time by sending a letter to the address below:

Mayo Clinic
Office for Human Research Protection
ATTN: Notice of Revocation of Authorization
201 Building 4-60
200 1st Street SW
Rochester, MN 55905

Alternatively, you may cancel your permission by emailing the Mayo Clinic Research Participant Advocate at: <a href="mailto:researchparticipantadvocate@mayo.edu">researchparticipantadvocate@mayo.edu</a>.

Please be sure to include in your letter or email:

- The name of the Principal Investigator,
- The study IRB number and /or study name, and
- Your contact information.

Your permission for Mayo Clinic to use and share your health information lasts until the end of this study, unless you cancel it. The study does not end until all data has been collected, checked (or audited), analyzed, and reported. Because research is an ongoing process, we cannot give you an exact date when the study will end. Sometimes this can be years after your study visits and/or activities have ended.

There is no expiration or end date related to the Sponsor's use of your health information received from Mayo Clinic as part of this study.

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34



#### Name and Clinic Number


# Frinted Name Person Obtaining Consent I have explained the research study to the participant. I have answered all questions about this research study to the best of my ability. Printed Name Date (mm/dd/yyyy) Time (hh:mm am/pm) Time (hh:mm am/pm) Time (hh:mm am/pm) Time (hh:mm am/pm)

IRB#: 18-003525 00 E-sign AS  IRB Doc. Ctrl # 10013.34